CLINICAL TRIAL: NCT05508776
Title: Interventional, Randomised, Partially Double-blind, Crossover, Positive-controlled, Single-dose Trial Investigating the Effect of LEO 152020 on Cardiac Repolarisation in Healthy Men and Women
Brief Title: A Trial to Evaluate the Effect of LEO 152020 on the Heart of Healthy People
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Collaborators: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LP0190-2212; U1111-1279-4625 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-08-18; First posted 2022-08-19 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Healthy Volunteers; Cardiac Repolarisation
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LEO 152020 Dose A (Experimental): A single oral dose of LEO 152020 Dose A according to the randomization schedule.
  Interventions: Drug: LEO 152020
- LEO 152020 Dose B (Experimental): A single dose of LEO 152020 Dose B according to the randomization schedule.
  Interventions: Drug: LEO 152020
- Moxifloxacin (Active Comparator): A single oral dose of moxifloxacin 400 mg according to the randomization schedule.
  Interventions: Drug: Moxifloxacin
- Placebo (Placebo Comparator): A single dose of placebo according to the randomization schedule.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LEO 152020 — Film-coated tablet
  Route of administration: Orally
  50 mg tablets
  Arms: LEO 152020 Dose A; LEO 152020 Dose B
Drug: Moxifloxacin — Tablet (may be film-coated depending on brand)
  Route of administration: Orally
  400 mg tablet
  Arms: Moxifloxacin
Drug: Placebo — Film-coated tablet
  Route of administration: Orally
  No active ingredient
  Arms: Placebo

SUMMARY:
The trial medicine (LEO 152020) is being developed to treat people with eczema.

The aims of this trial are to find out about:

* How the trial medicine affects participant's heart rhythm.
* How much of the trial medicine is absorbed into the bloodstream, and how quickly the body gets rid of it.
* The safety of the trial medicine and any side effects that might be related to it.

The trial will last up to 45 days, and there will be up to 6 visits.

Four treatment periods are planned for this trial. In each treatment period, participant will receive a single dose of the trial medicine at dose A, trial medicine at dose B, dummy tablet, or an approved medication named moxifloxacin (used for the treatment of bacterial infections). The order of these 4 treatment periods is chosen at random. Participant will receive all 4 treatments; it is only the order of the treatments that is random.

There will be 6 trial visits and they will include 1 screening visit, 4 treatment period visits and 1 final, follow-up visit at the clinic. The 4 treatment period visits will last for 3 days, from Day -1 (check-in to the clinic) to Day 2 (check-out of the clinic). There will be a period of at least 3 days between the 4 dosing occasions.

ELIGIBILITY:
Inclusion Criteria:

* Men or women between 18 and 55 years of age, inclusive, at screening.
* Body mass index between 18.0 and 30.0 kg/m2, inclusive.
* In good health at screening and check-in (as applicable) for Treatment Period 1, as assessed by the investigator (or designee) based on medical history, physical examination, 12-lead ECG, vital signs measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [e.g. suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable).
* Female subjects of childbearing potential must be willing to comply with the contraception requirements.

Exclusion Criteria:

* ECG with any clinically relevant abnormality, such as QTcF >450 ms (males) or >460 ms (females), QRS duration >110 ms, or PR interval >220 ms.
* Subjects at risk for Torsades de pointes based on any of the following:

  1. Uncorrected hypokalaemia or hypomagnesaemia at screening or check-in for Treatment Period 1, history of cardiac failure, history of clinically significant/symptomatic bradycardia.
  2. (Congenital) long QT syndrome or family history of idiopathic sudden death.
* Known history of ventricular arrhythmias.
* Second- or third-degree atrioventricular block.
* Use or intend to use any medications or products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to check-in for Treatment Period 1, considered to potentially impact subject safety or the objectives of the trial, as determined by the investigator (or designee).
* Use of tobacco- or nicotine-containing products within 3 months prior to check-in for Treatment Period 1, or positive cotinine at screening or check-in for Treatment Period 1.

Other protocol defined criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2022-09-16 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
Placebo-corrected change from baseline of LEO 152020 using QT interval corrected using Fridericia's formula (ΔΔQTcF) | Predose up to 24 hours postdose for each applicable treatment

SECONDARY OUTCOMES:
Change from baseline of Heart Rate (ΔHR) | Predose up to 24 hours postdose for each applicable treatment
  A continuous 12-lead electrocardiogram recording (Holter) will be performed for at least 25 hours, starting 1 hour predose on Day 1 and encompassing the entire period from prior to the first (predose) extraction time point until after the last (24 hours postdose) extraction time point.
Change from baseline of QT interval corrected using Fridericia's formula (ΔQTcF) | Predose up to 24 hours postdose for each applicable treatment
  A continuous 12-lead electrocardiogram recording (Holter) will be performed for at least 25 hours, starting 1 hour predose on Day 1 and encompassing the entire period from prior to the first (predose) extraction time point until after the last (24 hours postdose) extraction time point.
Change from baseline of Pulse Rate (ΔPR) | Predose up to 24 hours postdose for each applicable treatment
  A continuous 12-lead electrocardiogram recording (Holter) will be performed for at least 25 hours, starting 1 hour predose on Day 1 and encompassing the entire period from prior to the first (predose) extraction time point until after the last (24 hours postdose) extraction time point.
Change from baseline of QRS interval (ΔQRS) | Predose up to 24 hours postdose for each applicable treatment
  A continuous 12-lead electrocardiogram recording (Holter) will be performed for at least 25 hours, starting 1 hour predose on Day 1 and encompassing the entire period from prior to the first (predose) extraction time point until after the last (24 hours postdose) extraction time point.
Placebo-corrected, change from baseline of Heart Rate (ΔΔHR) | Predose up to 24 hours postdose for each applicable treatment
  A continuous 12-lead electrocardiogram recording (Holter) will be performed for at least 25 hours, starting 1 hour predose on Day 1 and encompassing the entire period from prior to the first (predose) extraction time point until after the last (24 hours postdose) extraction time point.
Placebo-corrected, change from baseline of Pulse Rate (ΔΔPR) | Predose up to 24 hours postdose for each applicable treatment
  A continuous 12-lead electrocardiogram recording (Holter) will be performed for at least 25 hours, starting 1 hour predose on Day 1 and encompassing the entire period from prior to the first (predose) extraction time point until after the last (24 hours postdose) extraction time point.
Placebo-corrected, change from baseline of QRS interval (ΔΔQRS) | Predose up to 24 hours postdose for each applicable treatment
  A continuous 12-lead electrocardiogram recording (Holter) will be performed for at least 25 hours, starting 1 hour predose on Day 1 and encompassing the entire period from prior to the first (predose) extraction time point until after the last (24 hours postdose) extraction time point.
Categorical outliers for QTcF, HR, PR interval, and QRS duration | Predose up to 24 hours postdose for each applicable treatment
  A continuous 12-lead electrocardiogram recording (Holter) will be performed for at least 25 hours, starting 1 hour predose on Day 1 and encompassing the entire period from prior to the first (predose) extraction time point until after the last (24 hours postdose) extraction time point.
Maximum observed plasma concentration of LEO 152020 (Cmax) | 0 to 24 hours postdose for each applicable treatment
Time to maximum plasma concentration of LEO 152020 (tmax) | 0 to 24 hours postdose for each applicable treatment
Area under the plasma concentration-time curve from time 0 to 24 hours postdose of LEO 152020 (AUC0-24). | 0 to 24 hours postdose for each applicable treatment
Area under the plasma concentration-time curve from time 0 to the time of last observed quantifiable concentration of LEO 152020 (AUC0-tlast) | 0 to 24 hours postdose for each applicable treatment
Area under the plasma concentration-time curve from time 0 extrapolated to infinity of LEO 152020 (AUC0-∞) | 0 to 24 hours postdose for each applicable treatment
Apparent terminal elimination half-life of LEO 152020 (t1/2) | 0 to 24 hours postdose for each applicable treatment
Apparent total plasma clearance of LEO 152020 (CL/F) | 0 to 24 hours postdose for each applicable treatment
Apparent volume of distribution during the terminal phase (Vz/F) | 0 to 24 hours postdose for each applicable treatment
Number of treatment-emergent adverse events (AEs) | Dosing on Day 1 of Treatment Period 1 to follow-up. (Up to 17 days)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (1):
- LEO Investigational Site, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Access Criteria: Data sharing is subject to approved scientifically sound research proposal and signed data agreement
URL: http://leopharmatrials.com/for-professionals